CLINICAL TRIAL: NCT03513263
Title: RCT: Evaluating the Effect of Oral Care for Periodontitis in Rhematoid Arthritis Patients in Uganda
Brief Title: Effect of Periodontal Care on Rhematoid Arthritis in Uganda
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SBS 457
Record Dates: First submitted 2018-03-16; First posted 2018-05-01 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-03

CONDITIONS: Rheumatoid Arthritis; Periodontal Diseases
MeSH Terms: conditions — Arthritis, Rheumatoid; Periodontal Diseases | interventions — Tooth Exfoliation

STUDY DESIGN:
Intervention Model Description: scaling and polishing plus oral hygiene instructions will be provided for the intervention arm while only oral hygiene instruction will be provided for the control arm. At the end of the six month follow up the control arm will also be provided with scaling and polishing.
Who Masked: Participant
Masking Description: the participants will not know the arm of the study they are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scaling and polishing plus oral hygiene instruction (Active Comparator): This arm will contain RA participants with PD who will continue with their treatment for RA and also receive the intervention of scaling and polishing plus oral hygiene instructions
  Interventions: Procedure: Scaling and polishing; Other: oral hygiene instructions
- only oral hygiene instructions (Sham Comparator): This arm will contain rheumatoid arthritis (RA) participants with periodontitis who will continue with their treatment for (RA) and also receive only oral hygiene instructions
  Interventions: Other: oral hygiene instructions

INTERVENTIONS:
Procedure: Scaling and polishing — An electronic scaler will be used to clean the gums
  Arms: Scaling and polishing plus oral hygiene instruction
Other: oral hygiene instructions — It will include 15-minute oral session with visual and verbal information on how to use a toothbrush, dental floss, and mouthwash correctly; how to clean bridges and dentures; and how and why to use a plaque disclosing test to perform tooth cleaning

SUMMARY:
this will be an RCT. to determine if non-surgical treatment for periodontitis can improve the disease activity score in 28 joints of rheumatoid arthritis in an African setting. Rheumatoid arthritis patients with periodontal disease will be randomised into an immediate intervention arm and a delayed intervention arm and both groups will be followed for two three monthly periods

DETAILED DESCRIPTION:
1. RESEARCH QUESTIONS

   * What is the prevalence of periodontitis among rthematoid arthritis patients attending the Mulago rheumatology clinic?
   * Does non-surgical treatment for periodontitis improve the disease activity score in 28 joints of rheumatoid arthritis in this local setting?
2. Problem statement It has been shown that intervention with nonsurgical treatment of periodontitis improved the periodontal condition of patients with periodontitis and RA, with beneficial effects upon the clinical and laboratory test parameters, disease activity scores in 28 joints (DAS28) and erythrocyte sedimentation rate (ESR). However, all the studies included in the reviews involved small samples sizes and follow-up periods of less than 6 months. And locally to our knowledge there is currently no published information looking at the role of periodontal disease among Ugandans with rheumatoid arthritis.
3. METHODS Objective 1 will be addressed with a cross sectional study design while objective 2 will be a randomized control intervention on a fresh sample of patients from the clinic who will be randomly assigned using computer generated random numbers.

Population : To address the objective 1 a total sample size of 146 randomly selected study participants.

For objective 2 the target sample size of 304 individuals or 152 individuals per group.

Procedures: On arrival to the dental clinic, the selected and previously consented participants will undergo a standardized interview. This will be followed by an oral examination to assess for: registration of plaque, bleeding on probing, probing depth and followed with the calculation of the Periodontal inflamed surface area score and clinical attachment loss, pick crevicular fluid using paper point for follow-up confirmatory polymerase chain reactions (PCR), quantification with quantitative real-time PCR (QPCR) experiments for P. gingivalis. At the end of the examination a peripheral blood sample will be obtained for: erythrocyte sedimentation rate to be factored in the determination of DAS 28 score. The remaining blood sample will be stored in the department of Anatomy for further studies latter pertaining to PD and RA.

Objective 2 RCT study Participants will be randomized into an immediate intervention arm and a delayed intervention arm.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older (of either gender).
2. RA diagnosed at least 2 year before V0.
3. DAS28 score between 3.2 and 5.1 during the month preceding V0.
4. No change in medication, dose, or formulation in RA treatment during the 3 months preceding V0.
5. Available for all study visits over 6 months
6. Presence of at least six natural teeth.
7. Ability to give written informed consent.
8. Having Periodontal Disease

Exclusion Criteria:

1. Chronic disorder requiring chronic or intermittent use of antibiotics.
2. Known hypersensitivity to chlorhexidine digluconate.
3. Participation in another intervention study.
4. Known contraindications to both amoxicillin and clindamycin.
5. Known contraindications to dental local anesthetic.
6. Pregnancy or lactation or intent to become pregnant

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
change in Disease Activity score of 28 joints | Two three monthly follow ups
  ≤ 3.2- inactive, >3.2 but ≤ 5.1 - moderate and > 5.1- very active

SECONDARY OUTCOMES:
change in clinical attachment loss | Two three monthly follow ups
  less than 2mm - improvement, more than 3 mm - getting worse

CONTACTS AND LOCATIONS:
Overall Officials: Ian Munabi, PhD, Study Director — MakCHS
Locations (1):
- Rheumatology clinic, medical outpatient department, Mulago national referral hospital and the Uganda, Kampala, Uganda